CLINICAL TRIAL: NCT07352345
Title: Head to Head, Prospective, Open Label Multicenter Study on the Diagnostic Efficacy of GPC3 Targeted PET Imaging and Enhanced Magnetic Resonance Imaging for Hepatocellular Carcinoma
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: XLan-251020
Record Dates: First submitted 2026-01-11; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Malignant Neoplasm of Liver
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PET imaging targeting GPC3 in hepatocellular carcinoma (Experimental): Determine if targeting GPC3 PET is safe and effective method for imaging of hepatocellular carcinoma
  Interventions: Drug: 68Ga-XH06

INTERVENTIONS:
Drug: 68Ga-XH06 — For Cancer patients, subjects should have targeting GPC3 scans.

SUMMARY:
This project intends to apply XH06 PET/CT or PET/MR imaging to patients suspected or diagnosed with hepatocellular carcinoma (liver mass), and compare it with enhanced magnetic resonance imaging. Using surgical/biopsy pathology as the gold standard, the diagnostic efficacy of XH06 PET/CT or PET/MR imaging for primary and metastatic lesions of hepatocellular carcinoma will be evaluated. The purpose is to further confirm the advantages of XH06 PET/CT or PET/MR in the diagnosis and staging of hepatocellular carcinoma through prospective, multicenter clinical studies, to compensate for the shortcomings of conventional imaging techniques in the diagnosis and staging of hepatocellular carcinoma, and to provide more accurate information to guide clinical treatment decisions for hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation and the patient or their legal representative is able to sign an informed consent form
2. Adult patients (aged 18 or above), regardless of gender 3: Patients with newly diagnosed hepatocellular carcinoma who are highly suspected or confirmed clinically (supporting evidence includes imaging data and histopathological examination, etc.) and agree to undergo histopathological examination (if not performed before imaging) 4: Patients with expected survival>3 months 5: Willing and able to follow schedule visits, treatment plans, laboratory and other relevant examinations

Exclusion Criteria:

* 1: Pregnant or lactating patients

  2: The patient or their legal representative is unable or unwilling to sign the informed consent form

  3: Acute systemic diseases and electrolyte imbalances

  4: Patients known to be allergic to XH06 imaging agent or synthetic excipients

  5: Individuals who are unable to complete PET/MR or PET/CT examinations (including inability to lie flat, claustrophobia, radiation phobia, etc.)

  6: Researchers believe that those with poor compliance or other factors that are not suitable for participating in this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Visual and standardized uptake values assessment of lesions and biodistribution | 1 year
  At least two experienced nuclear medicine physicians will conduct a visual analysis using consensus reading. The standardized uptake value (SUV) of tumor and organs will be measured after a semiquantitative analysis is conducted for each case. The SUV ranges from 0 to infinity, and a higher score means a higher uptake of targeting GPC3 nuclear probe by the tumor, which implies a greater threat of the tumor being malignant or higher stage.

SECONDARY OUTCOMES:
Pathological sections of tumour tissue | 1 year
  The excised tumour tissue was taken for immunohistochemistry to verify its GPC3 expression

CONTACTS AND LOCATIONS:
Locations (1):
- Wuhan union hosptital, Wuhan, Hubei, China